CLINICAL TRIAL: NCT07167849
Title: Optimizing a Digital Ultra-brief Treatment for Patients Waiting for Face-to-face Psychotherapy: An Investigation of Treatment Content, Human Support, and Patient Expectations (OPTIBRIEF)
Brief Title: Study on a Digital Ultra-Brief Intervention During Wait Times for Psychotherapy
Acronym: OPTIBRIEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2025-00844; HumRes67051 (Registry Identifier: HumRes); BASEC2025-00844 (Registry Identifier: BASEC); SNCTP000006475 (Registry Identifier: SNCTP)
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Depressive Disorders; Anxiety Disorders
Keywords: OPTIBRIEF; Ultra-brief treatment; Anxiety; Depression; Factorial trial; Wait time; Psychotherapy
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression

STUDY DESIGN:
Masking Description: Participants are assigned to 8 conditions. Due one factor being human support (on vs. off), that can reasonably be guessed, this is not considered full participant masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Problem-focused content (Experimental): Problem-focused condition of UKADO without human support or expectation fostering elements
  Interventions: Behavioral: UKADO Content - problem-focused
- Problem-focused content and expectation fostering elements (Experimental): Problem-focused condition of UKADO without human support but with expectation fostering elements
  Interventions: Behavioral: UKADO Content - problem-focused; Behavioral: Expectation fostering elements
- Problem-focused content and human support (Experimental): Problem-focused condition of UKADO with human support but no expectation fostering elements
  Interventions: Behavioral: UKADO Content - problem-focused; Behavioral: Human support
- Problem-focused content + human support + expectation fostering elements (Experimental): Problem-focused condition of UKADO with human support and expectation fostering elements
  Interventions: Behavioral: UKADO Content - problem-focused; Behavioral: Human support; Behavioral: Expectation fostering elements
- Resource-focused content (Experimental): Resource-focused condition of UKADO without human support and without expectation fostering elements
  Interventions: Behavioral: UKADO Content - resource-focused
- Resource-focused content and expectation fostering elements (Experimental): Resource-focused condition of UKADO without human support but with expectation fostering elements
  Interventions: Behavioral: UKADO Content - resource-focused; Behavioral: Expectation fostering elements
- Resource-focused content and human support (Experimental): Resource-focused condition of UKADO with human support but without expectation fostering elements
  Interventions: Behavioral: UKADO Content - resource-focused; Behavioral: Human support
- Resource-focused content + human support + expectation fostering elements (Experimental): Resource-focused condition of UKADO with human support and with expectation fostering elements
  Interventions: Behavioral: UKADO Content - resource-focused; Behavioral: Human support; Behavioral: Expectation fostering elements

INTERVENTIONS:
Behavioral: UKADO Content - problem-focused — UKADO is a digital ultra-brief intervention intended to reduce symptoms of depressive disorders and anxiety disorders. Content is either problem-focused or resource-focused. This version is problem-focused
  Arms: Problem-focused content; Problem-focused content + human support + expectation fostering elements; Problem-focused content and expectation fostering elements; Problem-focused content and human support
Behavioral: UKADO Content - resource-focused — UKADO is a digital ultra-brief intervention intended to reduce symptoms of depressive disorders and anxiety disorders. Content is either problem-focused or resource-focused. This version is resource-focused.
  Arms: Resource-focused content; Resource-focused content + human support + expectation fostering elements; Resource-focused content and expectation fostering elements; Resource-focused content and human support
Behavioral: Human support — Human support is provided as two weeks of guidance for study participants
  Arms: Problem-focused content + human support + expectation fostering elements; Problem-focused content and human support; Resource-focused content + human support + expectation fostering elements; Resource-focused content and human support
Behavioral: Expectation fostering elements — Patient in the expectation-fostering condition receive elements in UKADO that are meant to foster expectations.
  Arms: Problem-focused content + human support + expectation fostering elements; Problem-focused content and expectation fostering elements; Resource-focused content + human support + expectation fostering elements; Resource-focused content and expectation fostering elements

SUMMARY:
The OPTIBRIEF study investigates different versions of a digital ultra-brief intervention (UKADO - a German acronym for ultra-brief intervention against anxiety and depression online) during the waiting period for psychotherapy. Using a factorial trial design, the components 1) intervention content, 2) human support, and 3) expectation-fostering elements will be examined.

After completing initial questionnaires and participating in a diagnostic interview, participants are randomly assigned to one of eight groups and work through a specific version of UKADO. The program can be completed in a session of approximately 60 minutes, after which the exercises should continue to be used. Participants then complete another set of questionnaires at specific time points (after 2 weeks, 5 weeks, 9 weeks, and 24 weeks). A selection of participants also takes part in another telephone appointment to assess experiences with UKADO.

With the OPTIBRIEF study, the investigators aim to determine which version of the program is most suitable for individuals waiting for a psychotherapy slot. To this end, the investigators examine the effects on anxiety and depression symptom severity, as well as aspects such as participants' experiences with the program.

ELIGIBILITY:
Inclusion Criteria:

* Read the patient information and return signed written informed consent sheet
* Currently waiting for outpatient psychotherapy (self-report at baseline and assessed per telephone)
* Age ≥ 18 (self-report at baseline and assessed per telephone)
* Scoring equal to or above 10 on the PHQ-ADS (self-report at baseline)
* Fulfilling diagnostic criteria of one or more of the following disorders assessed with the Diagnostic Short-Interview for Mental Disorders (Mini-DIPS, DSM-5 version; Margraf et al., 2017): Major Depressive Disorder, Persistent Depressive Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, Generalized Anxiety Disorder
* Sufficient German skills (self-report at baseline)
* Access to the internet (self-report at baseline)

Exclusion Criteria:

* Acute suicidality assessed during the telephone interview (Mini-DIPS)
* Currently taking part in psychotherapy or a scheduled start of psychotherapy prior to the assessment 14 days post-randomization (assessed via self-report and during the DIPS telephone interview)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Depression and anxiety symptom severity assessed by the PHQ-ADS | At two weeks
  Self-reported depression and anxiety symptom severity will be measured using the Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS; Kroenke et al., 2016; 2019). The PHQ-ADS combines the Patient Health Questionnaire 9-item depression scale (PHQ-9) and 7-item Generalized Anxiety Disorder scale (GAD-7). Scores range from 0 to 48, with higher scores indicating greater symptom severity. The primary endpoint is at 2 weeks. Assessments will also be conducted at baseline, 5 weeks, 9 weeks, and 24 weeks.

SECONDARY OUTCOMES:
Depression and anxiety symptom severity assessed by the PHQ-ADS | 5 weeks, 9 weeks
  Self-reported depression and anxiety symptom severity will be measured using the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS; Kroenke et al., 2016; 2019). Scores range from 0 to 48, with higher scores indicating greater symptom severity. Assessments are conducted at baseline, 2 weeks, 5 weeks, 9 weeks, and 24 weeks.
Depression and anxiety symptom severity assessed by the PHQ-ADS | 24 weeks
  Self-reported depression and anxiety symptom severity will be measured using the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS; Kroenke et al., 2016; 2019). Scores range from 0 to 48, with higher scores indicating greater symptom severity. Assessments are conducted at baseline, 2 weeks, 5 weeks, 9 weeks, and 24 weeks.
Depression symptom severity | Baseline, 2 weeks, 5 weeks, 9 weeks, 24 weeks.
  Depressive symptoms assessed with the Patient Health Questionnaire-9 (PHQ-9) scale that is a part of the PHQ-ADS (Kroenke et al., 2016). The PHQ-9 measures the severity of depressive symptoms and has demonstrated high validity and reliability. Scores range from 0 (no depressive symptoms) to 27 (severe depressive symptoms).
Anxiety symptom severity | Baseline, 2 weeks, 5 weeks, 9 weeks, 24 weeks
  Anxiety symptoms assessed with the Generalized Anxiety Disorder-7 scale (GAD-7) that is a part of the PHQ-ADS (Kroenke et al., 2016). The GAD-7 measures the severity of generalized anxiety symptoms and has demonstrated strong validity and reliability. Scores range from 0 (no general anxiety symptoms) to 21 (severe general anxiety symptoms)
Quality of life (EQ-5D-5L) | Baseline, 2 weeks, 5 weeks, 9 weeks, 24 weeks
  Quality of life assessed with the European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L; Herdman et al., 2001). This measure includes five dimensions-Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression-each rated on a 5-point scale from 1 (no problems) to 5 (extreme problems).
Satisfaction with treatment | two weeks
  Satisfaction assessed with the Client Satisfaction Questionnaire-8 (CSQ-8; Attkisson & Zwick, 1982), adapted for internet interventions. The CSQ-8 consists of 8 items rated on a 4-point Likert scale, with higher scores indicating greater satisfaction. The German version has demonstrated high reliability and validity (Kriz et al., 2008).
Negative effects | 2 weeks, 5 weeks, 9 weeks, 24 weeks
  Negative treatment effects of UKADO assessed with the Negative Effects Questionnaire (NEQ; Rozental et al., 2019). This 20-item measure evaluates adverse effects during psychological treatments, including symptoms, therapy quality, dependency, stigma, and hopelessness.
Resource activation and problem mastery | 2 weeks, 5 weeks, 9 weeks
  Resource activation and problem mastery assessed with selected items from the Bern Post Session Report 2000, Patient and Therapist Versions (Flückiger et al., 2010), adapted for the digital intervention.
Therapeutic alliance | 2 weeks, 5 weeks, 9 weeks
  Therapeutic alliance measured with the Working Alliance Inventory for Guided Internet Interventions (WAI-I; Gomez Penedo et al., 2020), adapted to assess alliance with the study team. The 12 items assess agreement on therapeutic tasks, agreement on therapeutic goals, and emotional bond, rated on a 5-point Likert scale. Scores can range from 12 to 60, a higher score means a higher working alliance.
Treatment expectations | Baseline, two weeks, 5 weeks, 9 weeks
  Treatment expectations assessed with the Treatment Expectancy Questionnaire (TEX-Q; Alberts et al., 2020; Shedden-Mora et al., 2023), covering six subscales: Treatment benefit, Positive impact, Adverse events, Negative impact, Process, and Behavioral control. Scores range from 0 to 10, with higher scores indicating greater expectations.

OTHER OUTCOMES:
Patient experience interviews | 9 weeks
  Qualitative interviews conducted with a subset of participants using a study-specific guide developed to explore participants' experiences with the intervention.
Patient experience with UBT and its effect on f2f therapy experience at follow-up | 24 weeks
  Impact of UBT on f2f therapy experience (assessed with study-specific questions)
UBT uptake | 2 weeks
  Uptake of the UBT will be assessed at 2 weeks by reporting the number of patients who used the UBT (logged in).
UBT adherence | 2 weeks
  Usage of (adherence to) the UBT will be assessed at 2 weeks with a composite adherence score based on pages visited, time spent, and user input.
Psychotherapy uptake | 2 weeks, 5 weeks, 9 weeks, 24 weeks
  Self-reported psychotherapy uptake will be assessed via online questionnaires by recording the number of patients opting out of face-to-face (f2f) therapy after UBT and the number of patients who started f2f psychotherapy at each timepoint.
Psychotherapy use | 2 weeks, 5 weeks, 9 weeks, 24 weeks
  Self-reported psychotherapy use will be assessed via online questionnaire to record the number of sessions attended at each timepoint.
Adverse Events | Up to 24 weeks.
  The number and type of adverse events occurring during the study will be reported for the entire sample.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Luisa Bielinski, PhD, Principal Investigator — Department of Clinical Psychology and Psychotherpay, University of Bern
Locations (1):
- Department of Clinical Psychology and Psychotherapy, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol